CLINICAL TRIAL: NCT00121433
Title: The Role of Leptin in Modulating Vascular Tone and Endothelial Function in Obese and Normal Weight Adults: A Vascular-Protective Effect of Leptin?
Brief Title: Leptin and Endothelial Function
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Michigan (Other)
Collaborators: Amgen (Industry)
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: GCRC 1955; GCRC 1955; IRB 2003-0383
Record Dates: First submitted 2005-07-13; First posted 2005-07-21 (Estimated); Last update posted 2006-06-27 (Estimated); Status verified 2005-07

CONDITIONS: Healthy
MeSH Terms: interventions — Leptin

INTERVENTIONS:
Drug: leptin

SUMMARY:
The purpose of this trial was to determine if injections of leptin would improve vascular function in normal-weight, healthy volunteers.

DETAILED DESCRIPTION:
The researchers plan to enroll a total of 15 non-obese (BMI < 27 kg/m2) otherwise healthy adults into a randomized, double-blinded, cross-over study of the impact of recombinant methionyl human leptin 0.2 mg/kg SC, hereafter called rL, (Amgen Inc, Thousand Oaks, Calif) versus placebo SC (sorbitol and sodium acetate, pH 4.0 of same volume) in 15 non-obese adults. Subjects will have baseline vascular studies performed by brachial artery ultrasonography-flow-mediated dilatation and nitroglycerin mediated dilatation and blood drawn for measures of leptin levels. They will then receive rL SC or placebo SC (randomized order). They will then have vascular studies performed and blood levels drawn every 2 hours for 6 hours total. After completion of day 1, patients will return 1-4 weeks later and repeat the protocol crossed-over to the alternate intervention (rL or placebo).

ELIGIBILITY:
Inclusion Criteria:

* Healthy male or female ages 18-50.
* BMI < 27 kg/m2 for lean group

Exclusion Criteria:

* Any CVD risk factor (diabetes or fasting glucose > 126 mg/dL
* Hypertension or measured BP > 140/90 mmHg
* Current tobacco smoking within last month
* LDL>160 mg/dL, HDL<35 mg/dL)
* Renal insufficiency (creatinine > 1.4 mg/dL)
* Thyroid abnormalities (abnormal TSH)
* Established CVD (any atherosclerosis, or history of peripheral arterial disease, previous stroke, myocardial infarction, angina, heart failure, aortic aneurysms)
* Usage of medications which impact endothelial function within last month (folate, fish oil, Vitamin C or E, L-arginine, blood pressure or lipid-lowering medications, diabetes medications)

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 15
Dates: Start 2004-09; Study Completion 2004-12

PRIMARY OUTCOMES:
flow-mediated dilatation (FMD) of the brachial artery (conduit artery shear stress-mediated endothelial-dependent vasodilatation)

SECONDARY OUTCOMES:
basal brachial arterial diameter (BAD) (resting conduit artery tone)
basal brachial arterial blood flow (BABF) (resting resistance artery tone)